CLINICAL TRIAL: NCT06864754
Title: WashU DIEP Flap Video and Patient Understanding Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202503134
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Pre-operative anxiety; Patient understanding; Breast reconstruction; DIEP flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WashU DIEP Flap Video (Experimental): At the pre-operative appointment, patients will complete the pre-video survey (~10min) via RedCap, watch the video (~5min), and complete the post-video survey (~10min) via RedCap. During the standard of care follow-up appointment ≤ 30 days after surgery, consented patients will fill out a third survey via RedCap (~5min).
  Interventions: Other: WashU DIEP Flap Video

INTERVENTIONS:
Other: WashU DIEP Flap Video — Video uses visual cues and graphics to help explain complex procedures in a simplified, comprehensible fashion to patients.

SUMMARY:
Patients will complete a survey before and after watching the WashU DIEP Flap Video at their pre-operative standard of care visit, and a third survey at their post-operative standard of care visit. These surveys will use questions from SILS, APAIS, PEMAT, and AIM/IAM to assess the patient's health literacy, demographics questions, and questions concerning patient understanding and anxiety surrounding the procedure. The purpose of the post-op survey will be to assess how well the video set expectations of the procedure and recovery process and will repeat questions asked pre-operatively. Survey responses will be analyzed to determine if there are beneficial trends and improvement in patient understanding and anxiety due to adjunct video usage.

Primary Objective: The primary aim of the study is to determine if our animated video affects understanding and anxiety survey scores in patients undergoing DIEP breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to have DIEP-flap breast reconstruction at Barnes Jewish Hospital
* Speak English
* ≥ 18 years of age

Exclusion Criteria:

* Non-English speaking are excluded as the consent, questionnaires, and video are only available in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in understanding as measured by the Comprehension Assessment | Before video at pre-operative visit, after video at pre-operative visit, and at post-operative visit (estimated to be 3 months)
  The pre-op, pre-video survey includes a 10-question comprehension assessment. The pre-op, post-video survey repeats the comprehension assessment. Scores of the comprehension assessment will be compared before and after video watching per patient to determine change in understanding due to the video. It will be scored on a 10-point scale based on correct answers with a higher score meaning greater understanding of the procedure.
Change in anxiety as measured by the Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Before video at pre-operative visit, after video at pre-operative visit, and at post-operative visit (estimated to be 3 months)
  Scores of the APAIS will be compared before and after video watching per patient to determine change in anxiety due to the video. Scoring of APAIS will be per the literature (6-30 with higher score meaning greater anxiety).

SECONDARY OUTCOMES:
Appropriate expectation setting as measured by The Patient Education Materials Assessment Tool (PEMAT) | Before video at pre-operative visit and at post-operative visit (estimated to be 3 months)
  Will be used to assess video quality. Validated scoring will be used (0-12 with higher score meaning better quality).
Appropriate expectation setting as measured by the Acceptability of Intervention Measure (AIM) | At post-operative visit (estimated to be at 3 months)
  Validated survey which will be used per published scoring guidelines (8-40 with higher score meaning greater acceptability.
Appropriate expectation setting as measured by the Intervention Appropriateness Measure (IAM) | At post-operative visit (estimated to be at 3 months)
  Validated survey which will be used per published scoring guidelines (8-40 with higher score meaning greater appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Justin M Sacks, M.D., MBA, FACS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu